CLINICAL TRIAL: NCT02487381
Title: Gene-Environment-Interaction: Influence of the COMT Genotype on the Effects of Different Cannabinoids on the Endocannabinoid System, Cognition and Neuronal Oscillations
Brief Title: Gene-Environment-Interaction: Influence of the COMT Genotype on the Effects of Different Cannabinoids
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Principal Investigator, F Markus Leweke, Prof. Dr. F. Markus Leweke, Central Institute of Mental Health, Mannheim
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GEI-TCP II
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Healthy; Modeling Psychosis
Keywords: delta-9-tetrahydrocannabinol; cannabidiol; COMT; Volunteers
MeSH Terms: interventions — Dronabinol; Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- THC (Experimental): Subjects receive 20 mg delta-9-tetrahydrocannabinol (2 capsules containing 10 mg each) and corresponding cannabidiol placebo capsules.
  Interventions: Drug: delta-9-tetrahydrocannabinol; Drug: Placebo
- CBD (Experimental): Subjects receive 800 mg cannabidiol (4 capsules containing 200 mg each) and corresponding delta-9-tetrahydrocannabinol placebo capsules.
  Interventions: Drug: Cannabidiol; Drug: Placebo
- CBD+THC (Experimental): Subjects receive 800 mg cannabidiol (4 capsules containing 200 mg each) and 20 mg delta-9-tetrahydrocannabinol (2 capsules containing 10 mg each) a
  Interventions: Drug: delta-9-tetrahydrocannabinol; Drug: Cannabidiol
- Placebo (Placebo Comparator): Subjects receive corresponding delta-9-tetrahydrocannabinol and cannabidiol placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: delta-9-tetrahydrocannabinol
  Other Names: Dronabinol
  Arms: CBD+THC; THC
Drug: Cannabidiol
  Arms: CBD; CBD+THC
Drug: Placebo
  Arms: CBD; Placebo; THC

SUMMARY:
The study evaluates the gene-environment interaction of the COMT-genotype on the effects of the phytocannabinoids delta-9-tetrahydrocannabinol, cannabidiol or a combination of both on induction of psychotic symptoms, endocannabinoid levels in human body fluids, neuronal processing, and neural oscillations. In addition the effects of the phytocannabinoids on lipid levels in serum and cerebrospinal fluid, cognition, neural synchrony and neuronal processing assessed by EEG and fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent given by the subject
* Healthy young man (age between 18 and 45) insightful to the study (WST> 95)
* Right handedness
* At least one time consumption of Cannabis but less than 10 times/ per lifetime, no consumption of other psychotropic agents (despite coffee or nicotine), no alcohol abuse
* Negative drug-screening at the time of screening
* Body Mass Index between 18 and 30

Exclusion Criteria:

* Lack of accountability
* Participation in other interventional trials
* Severe medical or neurological illness, especially cardiovascular, renal, advanced respiratory, hematological or endocrinological failures or infectious diseases (acute hepatitis A, B or C or HIV) assessed at the time of the screening by the subject's history, clinical examination and laboratory testing, at the discretion of the investigator
* Any known psychiatric illness in the participant's history
* Known family history concerning psychiatric disorders
* Cannabis consumption within the last six months
* Consumption of any illegal drugs (except cannabis in history, see above)
* Intake of interfering medication, at the discretion of the investigator
* High intracranial pressure
* Any disorders in stereoscopic vision (measured by the TNO-Test, Lamerics, Utrecht) or hearing deficits
* Contraindications due to the Investigators Brochure Contraindication for Magnetic Resonance Imaging (e.g. cardiac pacemaker, claustrophobia, attached brace, in body metal, tattoos) or lumbar puncture (e.g. local or systemic infection, disturbance of blood coagulation, medication with anticoagulants like Phenprocoumon)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Syndrome Scale total score (PANSS T) from baseline to post drug intake of both on induction of psychotic symptoms, endocannabinoid levels in human body fluids, neuronal processing, and neural synchrony. | up to 4 hours

SECONDARY OUTCOMES:
Change in Positive and Negative Syndrome Scale (PANSS) subscores and clusters (baseline to post drug intake) | up to 4 hours
Change in neuropsychological parameters | up to 6 hours
Assessment of hallucinogen states (APZ) (post drug intake) | 1 day
Safety and tolerability assessments including (S)AEs, physical examination, vital signs (including heart rate and systolic and diastolic blood pressure in both supine and standing positions), and detailed laboratory assessments | 1 day
Metabolic markers post drug intake (blood) | up to 4 hours
Metabolic markers post drug intake (cerebrospinal fluid) | up to 4 hours
Neural synchrony and event-related potentials post drug intake | up to 5 hours

OTHER OUTCOMES:
Assessment of biomarker profiles in serum and cerebrospinal fluid of subjects. | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Central Institute of Mental Health, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Woelfl T, Rohleder C, Mueller JK, Lange B, Reuter A, Schmidt AM, Koethe D, Hellmich M, Leweke FM. Effects of Cannabidiol and Delta-9-Tetrahydrocannabinol on Emotion, Cognition, and Attention: A Double-Blind, Placebo-Controlled, Randomized Experimental Trial in Healthy Volunteers. Front Psychiatry. 2020 Nov 13;11:576877. doi: 10.3389/fpsyt.2020.576877. eCollection 2020. PMID 33304282